CLINICAL TRIAL: NCT01697956
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 6-Week Study Designed to Investigate the Effects of BDP Nasal Aerosol on the Hypothalamic-Pituitary-Adrenal (HPA)-Axis in Pediatric Subjects (6 to 11 Years of Age) With Perennial Allergic Rhinitis (PAR)
Brief Title: Hypothalamic-Pituitary-Adrenal (HPA)-Axis Study in Pediatric Subjects With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-AR-307
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Rhinitis
Keywords: Pediatric Subjects
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP Nasal Aerosol 80 mcg/day (Experimental): BDP nasal aerosol: 80 mcg dose once daily in the morning. Participants/parents administer 40 mcg BDP (one spray per nostril) during the 42 day (6 week) Treatment Period.
  Interventions: Drug: BDP
- Placebo Nasal Aerosol (Placebo Comparator): Participants/parents administer placebo (no medication) (one spray per nostril) once daily in the morning during the 42 day (6 week) Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BDP — Beclomethasone dipropionate (BDP) 80 mcg/day (40 mcg/spray, 1 spray/nostril, once daily - total 2 sprays/day) as a nasal aerosol.
  Other Names: QNASL®; Beclomethasone dipropionate
  Arms: BDP Nasal Aerosol 80 mcg/day
Drug: Placebo — Placebo (1 spray/nostril, once daily - total 2 sprays/day) as a nasal aerosol.
  Arms: Placebo Nasal Aerosol

SUMMARY:
The purpose of this study is to compare the effect of 6 weeks of treatment with beclomethasone dipropionate (BDP) nasal aerosol versus placebo on HPA-axis function, as assessed by 24-hour serum cortisol weighted mean, and to evaluate the safety and tolerability of BDP nasal aerosol, in subjects 6 to 11 years of age with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/(assent - if applicable)
* Male or female subjects 6-11 years of age
* General good health
* A documented history of PAR to a relevant perennial allergen for a minimum of 12 months
* Other criteria apply

Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes
* Participation in any investigational drug study within the 30 days preceding the Screening Visit 1 (SV1)
* Previous participation in a BDP nasal aerosol study as a randomized subject
* A known hypersensitivity to any corticosteroid or any of the excipients in the study medication formulation
* History of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations
* History of a respiratory infection or disorder within the 14 days preceding the Screening Visit 1 (SV1)
* Use of any prohibited concomitant medications within the prescribed (per protocol) withdrawal periods prior to the Screening Visit 1 (SV1)
* Other criteria apply
* Current smoker or current user of tobacco products at any time during the study; history of smoking or use of tobacco products within the past year

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh K Tantry, Ph.D., Principal Investigator — Teva Branded Pharmaceutical Products R&D
Locations (6):
- United States (6):
  - Teva Investigational Site 10305, Long Beach, California
  - Teva Investigational Site 10304, Stockbridge, Georgia
  - Teva Investigational Site 10300, Plymouth, Minnesota
  - Teva Investigational Site 10302, Normal Square, Pennsylvania
  - Teva Investigational Site 10301, New Braunfels, Texas
  - Teva Investigational Site 10303, San Antonio, Texas

REFERENCES:
- [Derived] Hampel FC Jr, Nayak NA, Segall N, Small CJ, Li J, Tantry SK. No hypothalamic-pituitary-adrenal function effect with beclomethasone dipropionate nasal aerosol, based on 24-hour serum cortisol in pediatric allergic rhinitis. Ann Allergy Asthma Immunol. 2015 Aug;115(2):137-42. doi: 10.1016/j.anai.2015.05.019. PMID 26250771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 110 subjects were screened. Participants were randomly assigned to either BDP nasal aerosol (80 mcg/day) or placebo nasal aerosol in a 2:1 ratio.
Period: Overall Study
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Started | 67 (enrolled and randomized) | 32 (enrolled and randomized)
Per Protocol Population | 66 | 31
Completed | 66 | 31
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per Protocol (PP) population included all data from randomized subjects obtained prior to experiencing major protocol deviations
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol | Total
Number analyzed (Participants) | 66 | 31 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (1.54) | 8.5 (1.65) | 9.0 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 35 | 11 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  White | 48 | 24 | 72
  Black | 17 | 6 | 23
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 16 | 10 | 26
  Not Hispanic or Latino | 50 | 21 | 71
Weight [Mean (Standard Deviation); unit: kg] | 37.5 (12.84) | 34.9 (12.89) | 36.7 (12.85)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.8 (4.01) | 18.2 (3.66) | 18.6 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Expressed As A Ratio) In 24-Hr Serum Cortisol Weighted Mean Following 6 Weeks Of Treatment
Description: The serum cortisol weighted mean (0-t), calculated by dividing the area under the concentration-time curve (AUC) from time zero to the time of the last measurable value over the 24-hour period by the sample collection time interval, was determined for each participant at baseline and Week 6, and the ratio of Week 6 over baseline was derived.
Time Frame: Baseline (Day 1, -24, -22, -20, -16, -12, -8, and 0 hours prior to study medication), End of Treatment (Day 43, (Immediately prior to study medication administration (Hour 0) and at 2, 4, 8, 12, 16, and 24 hours after study medication administration)
Population: Per protocol (PP) population
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 66 | 31
ratio | 1.04 (1.037) | 1.10 (1.053)
Statistical Analysis 1: Comparison: BDP Nasal Aerosol 80 mcg/Day vs Placebo Nasal Aerosol; The standard deviation of the logarithmically transformed data on the change from baseline (expressed as a ratio) in 24-hr serum cortisol weighted mean is assumed to be 0.30. Using this standard deviation, 90 subjects (approximately 60 and 30 subjects in the BDP Nasal Aerosol and placebo groups, respectively) will yield approximately 90% power to demonstrate non-inferiority between BDP Nasal Aerosol and placebo, if there is no true difference between treatment groups; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the lower limit of the two-sided 95% CI for the geometric mean ratio of BDP nasal aerosol versus placebo was greater than 0.80; ratio of BDP nasal aerosol to placebo = 0.91, 95% CI 2-sided [0.81 to 1.03]

2. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-t ) for Beclomethasone-17-monopropionate (17-BMP) and Beclomethasone Dipropionate (BDP)
Description: Beclomethasone-17-monopropionate (17-BMP) is the active metabolite of BDP. Plasma concentrations of 17-BMP or BDP that were below the lower-limit-of-quantitation (LLOQ), 20 or 10 pg/mL, respectively, were assigned a zero value when calculating descriptive statistics.
Time Frame: Day 42 (Predose (within 30 minutes prior to dose administration) and at 0.25 (15 min), 0.5 (30 min), 1, 1.5, 3, 6, 12, and 24 hours after final study medication administration)
Population: Per protocol population of participants administered BDP nasal aerosol 80 mcg/day
Measure: Mean (Standard Deviation); unit: h*pg/mL
Groups:
- 17-BMP Pharmacokinetic Parameters: PK values characterizing the active metabolite for BDP
- BDP Pharmacokinetic Parameters: PK values characterizing beclomethasone dipropionate (BDP)
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 66 | 66
h*pg/mL | 573.81 (508.727) | 45.60 (59.037)

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC0-24) for Beclomethasone-17-monopropionate (17-BMP) and Beclomethasone Dipropionate (BDP)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Per protocol population of participants administered BDP nasal aerosol 80 mcg/day. Plasma BDP concentrations were generally low and were only measurable over a short period of time.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 47 | 4
h*pg/mL | 619.06 (416.035) | 200.80 (69.939)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Beclomethasone-17-monopropionate (17-BMP) and Beclomethasone Dipropionate (BDP)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Per protocol population of participants administered BDP nasal aerosol 80 mcg/day.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 66 | 66
pg/mL | 142.68 (77.728) | 44.65 (36.454)

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for Beclomethasone-17-monopropionate (17-BMP) and Beclomethasone Dipropionate (BDP)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 66 | 58
hours | 1.15 (1.189) | 1.26 (3.590)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz ) for Beclomethasone-17-monopropionate (17-BMP)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Per protocol population of participants administered BDP nasal aerosol 80 mcg/day. Due to the short duration of measurable BDP concentrations in plasma, λz for BDP could not be estimated for any participants.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 45 | 0
1/hour | 0.31 (0.151) |

7. Secondary Outcome: Terminal Elimination Half-life (t1/2) for Beclomethasone-17-monopropionate (17-BMP)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Per protocol population of participants administered BDP nasal aerosol 80 mcg/day. Due to the short duration of measurable BDP concentrations in plasma, t1/2 for BDP could not be estimated for any participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 17-BMP Pharmacokinetic Parameters | BDP Pharmacokinetic Parameters
Number analyzed (Participants) | 45 | 0
hours | 3.10 (2.518) |

8. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (AEs)
Description: The intensity or severity of the AE was characterized as mild (AE which is easily tolerated), moderate (AE sufficiently discomforting to interfere with daily activity) or severe (AE which prevents normal daily activities).
  The causal relationship was characterized as not related (no reasonable possibility that the AE was caused by or attributed to the investigational product) or related reasonable possibility that the AE was caused by or attributed to the investigational product / a causal relationship cannot be ruled out).
  An SAE was defined as an AE that resulted in any of the following:
  * Death
  * Life-threatening
  * Required hospitalization or prolonged existing hospitalization
  * Persistent or significant disability or incapacity
  * A congenital abnormality or birth defect
  * An important medical event which required medical intervention to prevent any of the above outcomes.
Time Frame: Day 1- week 10
Population: Safety population which included all randomized participants who received at least one dose of randomized study medication.
Measure: Number; unit: participants
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Number analyzed (Participants) | 67 | 32
participants
  >=1 AEs | 22 | 13
  Withdrawn due to AEs | 0 | 0
  Severe AEs | 2 | 1
  Treatment-related AEs | 2 | 1
  >=1 SAEs | 0 | 0

9. Secondary Outcome: Participants With Shifts in Hematology Results From Normal at Screening to High or Low at End of Study
Description: Shifting to 'High' refers to starting the study within normal range and being outside the high-end of normal by end of study. Conversely, shifting to 'Low' refers to starting the study within normal range and being outside the low-end of normal by end of study.
  MCHC = mean corpuscular hemoglobin concentration MCV = mean corpuscular volume, or mean cell volume MCH = mean corpuscular hemoglobin or mean cell hemoglobin
Time Frame: Screening (Day -21 to -7), End of Study (Day 42)
Population: Safety population
Measure: Number; unit: participants
Groups:
- BDP Nasal Aerosol 80 mcg/Day - Shift to High; BDP Nasal Aerosol 80 mcg/Day - Shift to Low: BDP nasal aerosol: 80 mcg dose once daily in the morning. Participants/parents administer 40 mcg BDP (one spray per nostril) during the 42 day (6 week) Treatment Period.
- Placebo Nasal Aerosol - Shift to High; Placebo Nasal Aerosol - Shift to Low: Participants/parents administer placebo (no medication) (one spray per nostril) once daily in the morning during the 42 day (6 week) Treatment Period.
Arm/Group | BDP Nasal Aerosol 80 mcg/Day - Shift to High | BDP Nasal Aerosol 80 mcg/Day - Shift to Low | Placebo Nasal Aerosol - Shift to High | Placebo Nasal Aerosol - Shift to Low
Number analyzed (Participants) | 67 | 67 | 32 | 32
participants
  Hemaglobin (g/L) | 0 | 1 | 0 | 0
  Hematocrit (l/l) | 0 | 4 | 1 | 2
  MCHC (g/L) | 0 | 0 | 0 | 0
  MCV (FL) | 0 | 0 | 0 | 0
  MCH (pg) | 0 | 0 | 0 | 0
  Red blood cells (10^12/L) | 0 | 3 | 0 | 2
  Platelets (10^9/L) | 0 | 1 | 0 | 0
  White blood cells (10^9/L) | 0 | 9 | 0 | 2
  Basophils (10^9/L) | 0 | 0 | 0 | 0
  Eosinsphils (10^9/L) | 2 | 8 | 3 | 2
  Lymphocytes (10^9/L) | 0 | 1 | 0 | 1
  Monocytes (10^9/L) | 0 | 10 | 0 | 5
  Neutrophils (10^9/L) | 0 | 8 | 0 | 4
  Segmented neutrophils (10^9/L) | 0 | 8 | 0 | 4

10. Secondary Outcome: Participants With Shifts in Serum Chemistry Results From Normal at Screening to High or Low at End of Study
Description: Shifting to 'High' refers to starting the study within normal range and being outside the high-end of normal by end of study. Conversely, shifting to 'Low' refers to starting the study within normal range and being outside the low-end of normal by end of study.
  BUN = blood urea nitrogen AST = aspartate transaminase ALT = alanine transaminase GGT = gamma-glutamyl transpeptidase
Time Frame: Screening (Day -21 to -7), End of Study (Day 42)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | BDP Nasal Aerosol 80 mcg/Day - Shift to High | BDP Nasal Aerosol 80 mcg/Day - Shift to Low | Placebo Nasal Aerosol - Shift to High | Placebo Nasal Aerosol - Shift to Low
Number analyzed (Participants) | 67 | 67 | 32 | 32
participants
  Sodium (mmol/L) | 0 | 0 | 0 | 0
  Potassium (mmol/L) | 0 | 0 | 0 | 0
  Chloride (mmol/L) | 2 | 0 | 1 | 0
  Bicarbonate (mmol/L) | 0 | 8 | 0 | 3
  Glucose (mmol/L) | 1 | 1 | 1 | 2
  BUN (mmol/L) | 0 | 0 | 0 | 0
  Creatinine (micromol/L) | 0 | 0 | 0 | 1
  Calcium (mmol/L) | 1 | 0 | 0 | 0
  Phosphorus (mmol/L) | 0 | 0 | 0 | 0
  Total protein (g/L) | 0 | 0 | 0 | 0
  Albumin (g/L) | 0 | 0 | 0 | 0
  Uric acid (micromol/L) | 0 | 1 | 0 | 0
  AST (u/L) | 1 | 0 | 0 | 0
  ALT (u/L) | 0 | 0 | 0 | 0
  Alkaline phosphatase (u/L) | 0 | 0 | 0 | 0
  GGT (u/L) | 0 | 0 | 0 | 0
  Total bilirubin (micromol/L) | 0 | 0 | 0 | 0
  Lactate dehydrogenase (u/L) | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 10
Arm/Group | BDP Nasal Aerosol 80 mcg/Day | Placebo Nasal Aerosol
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/32
Other Adverse Events (participants affected / at risk) | 11/67 | 6/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP Nasal Aerosol 80 mcg/Day (N=67) | Placebo Nasal Aerosol (N=32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pyrexia (General disorders) | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.